CLINICAL TRIAL: NCT03493854
Title: A Phase III, Randomized, Multicenter, Open-Label, Two-Arm Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Subcutaneous Administration of the Fixed-Dose Combination of Pertuzumab and Trastuzumab in Combination With Chemotherapy in Patients With HER2-Positive Early Breast Cancer
Brief Title: A Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Subcutaneous Administration of the Fixed-Dose Combination of Pertuzumab and Trastuzumab in Combination With Chemotherapy in Participants With HER2-Positive Early Breast Cancer
Acronym: FeDeriCa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO40324; 2017-004897-32 (EudraCT Number)
Expanded Access: NCT04395508 (Approved for marketing)
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Results first posted 2020-06-25 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Docetaxel; Paclitaxel; pertuzumab; Trastuzumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy (Active Comparator): Participants will receive 8 cycles of investigator's choice of neoadjuvant chemotherapy. This will include either: 1) 4 cycles of dose-dense doxorubicin plus cyclophosphamide (ddAC) once every 2 weeks (Q2W) (given with granulocyte colony-stimulating factor [G-CSF] support as needed according to local guidelines) followed by paclitaxel Q1W for 12 weeks; or 2) 4 cycles of doxorubicin plus cyclophosphamide (AC) once every 3 weeks (Q3W) followed by docetaxel Q3W for 4 cycles. Pertuzumab and trastuzumab will be given intravenously (IV) for 4 cycles Q3W concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants will undergo surgery. Thereafter, participants will receive an additional 14 cycles of pertuzumab IV and trastuzumab IV for a total of 18 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Docetaxel; Drug: Paclitaxel; Drug: Pertuzumab IV; Drug: Trastuzumab IV; Drug: Trastuzumab SC; Procedure: Surgery; Radiation: Post-operative Radiotherapy; Drug: Hormone Therapy
- Arm B: FDC of Pertuzumab and Trastuzumab SC + Chemotherapy (Experimental): Participants will receive 8 cycles of investigator's choice of neoadjuvant chemotherapy. This will include either: 1) 4 cycles of ddAC Q2W (given with G-CSF support as needed according to local guidelines) followed by paclitaxel once every week (QW) for 12 weeks; or 2) 4 cycles of AC Q3W followed by docetaxel Q3W for 4 cycles. The fixed-dose combination (FDC) of pertuzumab and trastuzumab will be given subcutaneously (SC) for 4 cycles (Q3W) concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants will undergo surgery. Thereafter, participants will receive an additional 14 cycles of the FDC of pertuzumab and trastuzumab SC for a total of 18 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Docetaxel; Drug: Paclitaxel; Drug: FDC of Pertuzumab and Trastuzumab SC; Procedure: Surgery; Radiation: Post-operative Radiotherapy; Drug: Hormone Therapy

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m2 will be administered IV on Day 1 of each cycle of treatment (as part of ddAC Q2W or AC Q3W) for Cycles 1-4.
Drug: Doxorubicin — Doxorubicin 60 mg/m2 will be administered IV on Day 1 of each cycle of treatment (as part of either ddAC Q2W or AC Q3W) for Cycles 1-4.
Drug: Docetaxel — As part of one of the two investigator's choices of chemotherapy (AC followed by docetaxel), docetaxel 75 mg/m2 will be administered IV on Day 1 of Cycle 5 and then 100 mg/m2 IV at the discretion of the investigator for Cycles 6-8 (Q3W), if no dose-limiting toxicity occurs.
Drug: Paclitaxel — As part of one of the two investigator's choices of chemotherapy (ddAC followed by paclitaxel), paclitaxel 80 mg/m2 will be administered IV QW for 12 weeks.
Drug: Pertuzumab IV — Pertuzumab will be administered as a fixed non-weight-based dose of 840-mg IV loading dose and then 420-mg IV maintenance dose Q3W.
  Other Names: Perjeta; RO4368451
  Arms: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy
Drug: FDC of Pertuzumab and Trastuzumab SC — The FDC of pertuzumab and trastuzumab will be administered SC at a fixed non-weight-based dose. A loading dose of 1200 mg SC pertuzumab and 600 mg SC trastuzumab is then followed by a maintenance dose of 600 mg SC pertuzumab and 600 mg SC trastuzumab Q3W.
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; RO7198574; RG6264
  Arms: Arm B: FDC of Pertuzumab and Trastuzumab SC + Chemotherapy
Drug: Trastuzumab IV — Trastuzumab will be administered as an 8-mg/kg IV loading dose and then 6 mg/kg IV maintenance dose Q3W.
  Other Names: Herceptin; RO0452317
  Arms: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy
Drug: Trastuzumab SC — After surgery (from Cycle 9 onwards), participants in Arm A will be allowed to switch from trastuzumab IV to trastuzumab SC, at the discretion of the investigator, in the countries where trastuzumab SC is routinely used. For participants who switch, a fixed dose of 600 mg trastuzumab SC (irrespective of the patient's weight) will be administered in the adjuvant phase.
  Other Names: Herceptin; RO0452317
  Arms: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy
Procedure: Surgery — Participants in both cohorts are scheduled to undergo surgery after 8 cycles of neoadjuvant therapy. Participants may undergo breast-conserving surgery or mastectomy according to routine clinical practice.
Radiation: Post-operative Radiotherapy — If indicated, radiotherapy is given after chemotherapy and surgery, during adjuvant HER2-targeted therapy and hormone therapy (for hormone-receptor positive disease).
Drug: Hormone Therapy — For hormone receptor positive breast cancer, tamoxifen or aromatase inhibitors will be allowed as adjuvant hormone therapy for postmenopausal participants and with ovarian suppression or ablation for premenopausal participants in countries where it has been registered for this indication. Its use must be consistent with the registered label. Hormone therapy is given after chemotherapy and surgery during adjuvant HER2-targeted therapy.

SUMMARY:
This is a global Phase III, two-arm, open-label, multicenter, randomized study to investigate the pharmacokinetics, efficacy, and safety of the fixed-dose combination (FDC) of pertuzumab and trastuzumab for subcutaneous (SC) administration in combination with chemotherapy in patients with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer in the neoadjuvant/adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
* Female and male patients with Stage II - IIIC (T2-T4 plus any N, or any T plus N1-N3, M0), locally advanced, inflammatory, or early-stage, unilateral, and histologically confirmed invasive breast cancer
* Primary tumor >2 cm in diameter, or node-positive disease (clinically or on imaging, and node positivity confirmed with cytology and/or histopathology)
* HER2-positive breast cancer confirmed by a central laboratory prior to study enrollment. HER2-positive status will be determined based on pretreatment breast biopsy material.
* Hormone receptor status of the primary tumor, centrally confirmed
* Patient agreement to undergo mastectomy or breast conserving surgery after neoadjuvant therapy
* Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue block for central confirmation of HER2 and hormone receptor status and additional biomarker research
* Baseline left ventricular ejection fraction (LVEF) ≥55% measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* For women of childbearing potential (WOCBP) who are sexually active: agreement to remain abstinent or use one highly effective non-hormonal contraceptive method with a failure rate of <1% per year, or two effective non-hormonal contraceptive methods during the treatment period and for 7 months after the last dose of HER2-targeted therapy, and agreement to refrain from donating eggs during this same period
* For men: men must remain abstinent or use a condom with a spermicidal product during the treatment period and for 7 months after the last dose of HER2-targeted therapy to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
* A negative serum pregnancy test must be available prior to randomization for WOCBP, unless they have undergone surgical sterilization
* No major surgical procedure unrelated to breast cancer within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment

Exclusion Criteria:

* Stage IV (metastatic) breast cancer
* Patients with a history of invasive breast cancer
* Patients with a history of concurrent or previously treated non-breast malignancies except for appropriately treated 1) non-melanoma skin cancer and/or 2) in situ carcinomas, including cervix, colon, and skin
* Patients who have received any previous systemic therapy for treatment or prevention of breast cancer, or radiation therapy for treatment of cancer
* Patients who have a past history of ductal carcinoma in situ or lobular carcinoma in situ if they have received any systemic therapy for its treatment or radiation therapy to the ipsilateral breast
* Patients with high-risk for breast cancer who have received chemo-preventative drugs in the past are not allowed to enter the study
* Patients with multicentric breast cancer, unless all tumors are HER2-positive
* Patients with bilateral breast cancer
* Patients who have undergone an excisional biopsy of primary tumor and/or axillary lymph nodes
* Axillary lymph node dissection prior to initiation of neoadjuvant therapy
* Sentinel lymph node biopsy prior to neoadjuvant therapy
* Treatment with any investigational drug within 28 days prior to randomization
* Serious cardiac illness or medical conditions
* Inadequate bone marrow function, renal function or impaired liver function
* Current severe, uncontrolled systemic disease that may interfere with planned treatment
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 7 months after the last dose of HER2-targeted therapy
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Known active liver disease, for example, active viral hepatitis infection, autoimmune hepatic disorders, or sclerosing cholangitis
* Concurrent, serious, uncontrolled infections, or known infection with HIV
* Known hypersensitivity to study drugs, excipients, and/or murine proteins
* Current chronic daily treatment with corticosteroids
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, colon, skin, and/or non-melanoma skin carcinoma
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease, coronary heart disease, clinically significant electrolyte abnormalities, or family history of sudden unexplained death or long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (107):
- United States (4):
  - Maryland Oncology Hematology, Rockville, Maryland
  - San Juan Oncology Associates, Farmington, New Mexico
  - Levine Cancer Institute, Charlotte, North Carolina
  - Northwest Medical Specialties, Lakewood, Washington
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - COIBA, Provincia de Buenos Aires
- Belgium (6):
  - Institut Jules Bordet, Anderlecht
  - GHdC Site Notre Dame, Charleroi
  - UZ Antwerpen, Edegem
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Ste-Elisabeth, Namur
- Brazil (3):
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Perola Byington, São Paulo, São Paulo
- Canada (5):
  - Royal Victoria Hospital, Barrie, Ontario
  - Lakeridge Health Center; R. S. MacLaughlin Durham Regional Cancer Center, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke - Hopital Fleurimont, Sherbrooke, Quebec
- Czechia (2):
  - Masarykuv onkologicky ustav, Brno
  - Multiscan s.r.o., Pardubice
- France (8):
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Institut Sainte Catherine, Avignon
  - CHRU Besançon, Besançon
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Curie; Oncologie Medicale, Paris
  - APHP - Hospital Saint Louis, Paris
  - ICO - Site René Gauducheau, Saint-Herblain
- Germany (8):
  - Klinikum Augsburg; Frauenklinik, Augsburg
  - Hochwaldkrankenhaus; Abt.Gynäkologie Geburtshilfe u.Senologie, Bad Nauheim
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - St. Johannes-Hospital, Dortmund
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - Gynäkologie Kompetenzzentrum; Praxis Dr. med. Carsten Hielscher, Stralsund
- Italy (6):
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE;U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Università degli Studi Federico II; Clinica di Oncologia Medica, Napoli, Campania
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Uni Degli Studi Di Genova ; Clinica Di Medicina Interna Ad Indirizzo Oncologico, Genoa, Liguria
  - ASST DI LECCO; Oncologia Medica, Lecco, Lombardy
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto
- Japan (16):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hyogo Medical University Hospital, Hyōgo
  - Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Fukushima Medical University Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - St. Luke's International Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Mexico (3):
  - Iem-Fucam, D.F., Mexico CITY (federal District)
  - Centro Médico Zambrano Hellion, Monterrey, Nuevo León
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
- Poland (6):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej - Curie, Bialystok
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice; Centr.Diagn.i Lecz.Chor.Piersi, Gliwice
  - Szpital Uniwersytecki w Krakowie; Oddzial Kliniczny Onkologii i Poradnia Onkologiczna, Krakow
  - Zachodniopomorskie Centrum Onkologii, Osrodek Innowacyjnosci, Rozwoju i Badan Klinicznych, Szczecin
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad; Klinika Nowtw.Piersi i Chir.Rekonstr, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Russia (6):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan', Tatarstan Republic
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Omsk Region Clinical Oncology Dispensary; 1St Sergical Department, Omsk
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (9):
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital de Cruces; Servicio de Oncología Médica, Barakaldo, Vizcaya
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Taiwan (3):
  - China Medical University Hospital; Surgery, Taichung
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - Chang Gung Medical Foundation - Linkou; Dept of Surgery, Taoyuan District
- Thailand (3):
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital; Department of Surgery/Head Neck and Breast Unit; Clinical Trial, Chiang Mai
  - Songklanagarind Hospital; Department of Surgery, Songkhla
- Ukraine (5):
  - Municipal Noncommercial Institution Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk
  - National Cancer Institute MOH of Ukraine, Kiev
  - Lviv State Oncology Regional Treatment and Diagnostic Centre, Lviv
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
- United Kingdom (7):
  - Brighton and Sussex Univ Hosp, Brighton
  - Velindre Cancer Centre, Cardiff
  - St Georges University Hospitals NHS Foundation Trust, London
  - Christie Hospital NHS Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Peterborough City Hospital, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical-trials/data-sharing/).

REFERENCES:
- [Derived] Tan AR, Im SA, Mattar A, Colomer R, Stroyakovskii D, Nowecki Z, De Laurentiis M, Pierga JY, Jung KH, Schem C, Hogea A, Badovinac Crnjevic T, Heeson S, Shivhare M, Kirschbrown WP, Restuccia E, Jackisch C; FeDeriCa study group. Fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection plus chemotherapy in HER2-positive early breast cancer (FeDeriCa): a randomised, open-label, multicentre, non-inferiority, phase 3 study. Lancet Oncol. 2021 Jan;22(1):85-97. doi: 10.1016/S1470-2045(20)30536-2. Epub 2020 Dec 21. PMID 33357420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 607 patients were screened, 500 of whom were randomized.
Groups:
- Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy: Participants received 8 cycles of investigator's choice of neoadjuvant chemotherapy. This included either: 1) 4 cycles of dose-dense doxorubicin plus cyclophosphamide (ddAC) once every 2 weeks (Q2W) (given with granulocyte colony-stimulating factor [G-CSF] support as needed according to local guidelines) followed by paclitaxel QW for 12 weeks; or 2) 4 cycles of doxorubicin plus cyclophosphamide (AC) once every 3 weeks (Q3W) followed by docetaxel Q3W for 4 cycles. Pertuzumab and trastuzumab were given intravenously (IV) for 4 cycles Q3W concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants underwent surgery. Thereafter, participants received an additional 14 cycles of pertuzumab IV and trastuzumab IV for a total of 18 (neo)adjuvant anti-HER2 treatment cycles.
- Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy: Participants received 8 cycles of investigator's choice of neoadjuvant chemotherapy. This included either: 1) 4 cycles of ddAC Q2W (given with G-CSF support as needed according to local guidelines) followed by paclitaxel once every week (QW) for 12 weeks; or 2) 4 cycles of AC Q3W followed by docetaxel Q3W for 4 cycles. The fixed-dose combination (FDC) of pertuzumab and trastuzumab was given subcutaneously (SC) for 4 cycles (Q3W) concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants underwent surgery. Thereafter, participants received an additional 14 cycles of the FDC of pertuzumab and trastuzumab SC for a total of 18 (neo)adjuvant anti-HER2 treatment cycles.
Period: Neoadjuvant Treatment Phase (24 Weeks)
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Started (Intent-to-Treat (ITT) Population) | 252 (This includes all randomized participants.) | 248 (This includes all randomized participants.)
Received at Least One Dose of Study Drug (Safety Population) | 252 | 248
Completed | 242 | 234
Not Completed | 10 | 14
Not completed — Adverse Event | 3 | 5
Not completed — Death | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Progressive Disease | 3 | 3
Not completed — Other | 1 | 2
Not completed — Other | 1 | 0
Period: Surgery & Adjuvant Treatment (42 Weeks)
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Started (Completed Neoadjuvant Treatment Phase) | 242 | 234
Completed Surgery | 239 | 234
Completed | 209 | 217
Not Completed | 33 | 17
Not completed — Adverse Event | 12 | 7
Not completed — Lack of Efficacy | 0 | 2
Not completed — Progressive Disease | 4 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Other | 7 | 2
Not completed — Death | 1 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Disease Relapse | 4 | 1
Period: Treatment-Free Follow-Up (up to 3 Years)
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Started | 247 (In addition to participants who completed the previous periods, those who prematurely withdrew from (neo)adjuvant treatment entered the follow-up phase.) | 241 (In addition to participants who completed the previous periods, those who prematurely withdrew from (neo)adjuvant treatment entered the follow-up phase.)
Completed | 223 | 219
Not Completed | 24 | 22
Not completed — Death | 10 | 11
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy: Participants received 8 cycles of investigator's choice of neoadjuvant chemotherapy. This included either: 1) 4 cycles of dose-dense doxorubicin plus cyclophosphamide (ddAC) once every 2 weeks (Q2W) (given with granulocyte colony-stimulating factor [G-CSF] support as needed according to local guidelines) followed by paclitaxel QW for 12 weeks; or 2) 4 cycles of doxorubicin plus cyclophosphamide (AC) once every 3 weeks (Q3W) followed by docetaxel Q3W for 4 cycles. Pertuzumab and trastuzumab were given intravenously (IV) for 4 cycles Q3W concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants underwent surgery. Thereafter, participants received an additional 14 cycles of pertuzumab IV and trastuzumab IV for a total of 18 cycles.
- Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy: Participants received 8 cycles of investigator's choice of neoadjuvant chemotherapy. This included either: 1) 4 cycles of ddAC Q2W (given with G-CSF support as needed according to local guidelines) followed by paclitaxel once every week (QW) for 12 weeks; or 2) 4 cycles of AC Q3W followed by docetaxel Q3W for 4 cycles. The fixed-dose combination (FDC) of pertuzumab and trastuzumab was given subcutaneously (SC) for 4 cycles (Q3W) concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants underwent surgery. Thereafter, participants received an additional 14 cycles of the FDC of pertuzumab and trastuzumab SC for a total of 18 cycles.
- Total: Total of all reporting groups
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy | Total
Number analyzed (Participants) | 252 | 248 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (10.8) | 51.7 (10.7) | 51.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 248 | 498
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 42 | 74
  Not Hispanic or Latino | 200 | 189 | 389
  Unknown or Not Reported | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 10 | 20
  Asian | 54 | 51 | 105
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 164 | 165 | 329
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 19 | 16 | 35
Randomization Stratification Factors: Hormone Receptor Status [Count of Participants; unit: Participants] — Hormone receptor status was based on central assessment of participant samples for estrogen receptor (ER) and progesterone receptor (PgR) negativity or positivity.
  Participants
    ER Negative and PgR Negative | 97 | 96 | 193
    ER Positive and PgR Positive | 155 | 151 | 306
    Unknown | 0 | 1 | 1
Randomization Stratification Factors: Clinical Stage at Presentation [Count of Participants; unit: Participants]
  Stage II-IIIA | 201 | 198 | 399
  Stage IIIB-IIIC | 51 | 50 | 101
Randomization Stratification Factors: Neoadjuvant Chemotherapy Regimen [Count of Participants; unit: Participants] — AC = doxorubicin plus cyclophosphamide; ddAC = dose-dense doxorubicin plus cyclophosphamide
  Participants
    ddAC Followed by Paclitaxel | 120 | 120 | 240
    AC Followed by Docetaxel | 132 | 128 | 260

OUTCOME MEASURES:

1. Primary Outcome: Trough Serum Concentration (Ctrough) of Pertuzumab During Cycle 7 (Pre-Dose Cycle 8)
Description: The observed pertuzumab trough serum concentration (Ctrough) at Cycle 7 was assessed following 3 cycles of pertuzumab IV and trastuzumab IV or the fixed-dose combination (FDC) of pertuzumab and trastuzumab SC. The Per Protocol Pharmacokinetics (PK) analysis population includes all enrolled participants who adhered to the protocol. Exclusions from the Per Protocol PK analysis population were made for the following reasons: participants were missing the Ctrough pre-dose Cycle 8 PK sample, participants with a Ctrough sample collected with at least 2 days deviation from the planned date on Day 21 (i.e., before Day 19 or after Day 23), participants given a dose amount that deviated from the planned dose by >20% within 3 cycles (from Cycle 5), participants with a dose delay of more than 7 days, a subcutaneous injection site other than thigh was used, if the Cycle 8 pre-dose and post-dose samples were switched, and an assay error impacting Ctrough measurement.
Time Frame: Pre-dose on Cycle 8, Day 1 (up to 21 weeks)
Population: Per Protocol PK Population: includes only participants who adhered to the pre-specified criteria for the schedule of pharmacokinetic assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 203 | 206
micrograms per millilitre (μg/mL) | 72.4 (34.1) | 88.7 (33.6)
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; The null hypothesis was that the pertuzumab Arm A SC dose is inferior to the pertuzumab Arm B IV dose (i.e., the CtroughSC/CtroughIV geometric mean ratio of the SC dose of pertuzumab relative to the IV dose is not greater than 0.8); Test type: Non-Inferiority — The null hypothesis could be rejected and non-inferiority concluded if the lower bound of the 90% confidence interval of the geometric mean ratio was ≥0.8; Geometric Mean Ratio = 1.22, 90% CI 2-sided [1.14 to 1.31] — The CtroughSC/CtroughIV geometric mean ratio was calculated as the SC dose of pertuzumab (Arm B) relative to the pertuzumab IV dose (Arm A)

2. Secondary Outcome: Ctrough of Trastuzumab During Cycle 7 (Pre-Dose Cycle 8)
Description: The observed trastuzumab trough serum concentration (Ctrough) at Cycle 7 was assessed following 3 cycles of pertuzumab IV and trastuzumab IV or the fixed-dose combination (FDC) of pertuzumab and trastuzumab SC. The Per Protocol Pharmacokinetics (PK) analysis population includes all enrolled participants who adhered to the protocol. Exclusions from the Per Protocol PK analysis population were made for the following reasons: participants were missing the Ctrough pre-dose Cycle 8 PK sample, participants with a Ctrough sample collected with at least 2 days deviation from the planned date on Day 21 (i.e., before Day 19 or after Day 23), participants given a dose amount that deviated from the planned dose by >20% within 3 cycles (from Cycle 5), participants with a dose delay of more than 7 days, a subcutaneous injection site other than thigh was used, if the Cycle 8 pre-dose and post-dose samples were switched, and an assay error impacting Ctrough measurement.
Time Frame: Pre-dose on Cycle 8, Day 1 (up to 21 weeks)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milllilitre (μg/mL)
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 203 | 206
micrograms per milllilitre (μg/mL) | 43.2 (34.7) | 57.5 (37.0)
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; The null hypothesis was that the trastuzumab Arm B SC dose is inferior to the Arm A trastuzumab IV dose (i.e., the CtroughSC/CtroughIV geometric mean ratio of the SC dose of trastuzumab relative to the IV dose is not greater than 0.8); Test type: Non-Inferiority — The null hypothesis could be rejected and non-inferiority concluded if the lower bound of the 90% confidence interval of the geometric mean ratio was ≥0.8. Non-inferiority was tested in hierarchical order after the primary outcome measure, to adjust for multiple statistical testing and control the type I error at one sided 5% significance level; Geometric Mean Ratio = 1.33, 90% CI 2-sided [1.24 to 1.43] — The CtroughSC/CtroughIV geometric mean ratio was calculated as the SC dose of trastuzumab (Arm B) relative to the trastuzumab IV dose (Arm A)

3. Secondary Outcome: Percentage of Participants With Total Pathological Complete Response (tpCR), According to Local Pathologist Assessment
Description: Total pCR (tpCR) was defined as eradication of invasive disease in the breast and axilla; that is, ypT0/is ypN0, according to the local pathologists' assessment. Pathologic response to therapy was determined at the time of surgery. The tpCR rate is the percentage of participants in the ITT population who achieved a tpCR. Participants with missing data for tpCR (i.e., do not undergo surgery or have an invalid pCR assessment) were included in the analysis and classified as non-responders. Rates of tpCR were calculated in each treatment arm and were assessed using the difference between the Arm B: Pertuzumab and Trastuzumab FDC SC and the Arm A: Pertuzumab IV and Trastuzumab IV tpCR rates and corresponding 95% Clopper-Pearson confidence intervals (CIs). The difference between the tpCR rates along with corresponding 95% Hauck-Anderson CIs were calculated. The lower bound of the CI will reliably reflect the largest tpCR difference that can be considered unlikely.
Time Frame: Following completion of surgery (up to 33 weeks)
Population: ITT Population: includes all enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Percentage of participants | 59.5 [53.2 to 65.6] | 59.7 [53.3 to 65.8]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only. tpCR was analyzed outside of a hypothesis-testing framework and according to the methodology outlined in the outcome measure description; Difference in tpCR Rate = 0.15, 95% CI 2-sided [-8.67 to 8.97] — Difference in tpCR rate was calculated as Arm B: PH FDC SC minus Arm A: P+H IV

4. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to Invasive Disease-Free Survival (iDFS; Excluding Second Primary Non-Breast Cancer [SPNBC]) Criteria
Description: iDFS (excluding SPNBC) is defined as the time from the first date of no disease (i.e., the date of primary surgery) to the first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence; ipsilateral local-regional invasive breast cancer reccurrence; distant recurrence; contralateral invasive breast cancer; or death attributable to any cause. Ipsilateral or contralateral in situ disease and SPNBC (including in situ carcinomas and non-melanoma skin cancers) will not be counted as progressive disease or relapse.
Time Frame: At 1, 2, 3, and 4 years
Population: The analysis population included all participants who had undergone surgery. The number analyzed at each landmark timepoint represents the number of participants who were remaining at risk for an event.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 239 | 234
Percentage of participants
  1 Year: number analyzed (Participants) | 219 | 222
  1 Year | 96.07 [93.55 to 98.59] | 97.37 [95.30 to 99.45]
  2 Years: number analyzed (Participants) | 208 | 205
  2 Years | 92.98 [89.66 to 96.30] | 90.75 [86.98 to 94.52]
  3 Years: number analyzed (Participants) | 194 | 199
  3 Years | 90.71 [86.93 to 94.50] | 89.86 [85.93 to 93.79]
  4 Years: number analyzed (Participants) | 31 | 23
  4 Years | 89.60 [85.54 to 93.65] | 88.50 [84.34 to 92.66]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only; p = 0.5216, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.68 to 2.11]

5. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to iDFS (Including SPNBC) Criteria
Description: Invasive disease-free survival (iDFS) including second primary non-breast cancer (SPNBC) is defined as the time from the first date of no disease (i.e., the date of primary surgery) to the first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence; ipsilateral local-regional invasive breast cancer reccurrence; distant recurrence; contralateral invasive breast cancer; or death attributable to any cause. It also includes SPNBC as an event (with the exception of non-melanoma skin cancers and in situ carcinoma of any site).
Time Frame: At 1, 2, 3, and 4 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 239 | 234
Percentage of participants
  1 Year: number analyzed (Participants) | 218 | 221
  1 Year | 95.63 [92.99 to 98.28] | 96.94 [94.70 to 99.17]
  2 Years: number analyzed (Participants) | 206 | 202
  2 Years | 92.10 [88.60 to 95.60] | 89.44 [85.44 to 93.43]
  3 Years: number analyzed (Participants) | 191 | 196
  3 Years | 89.39 [85.37 to 93.40] | 88.54 [84.40 to 92.69]
  4 Years: number analyzed (Participants) | 31 | 23
  4 Years | 88.27 [84.01 to 92.53] | 87.64 [83.35 to 91.93]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only; p = 0.5992, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.68 to 1.97]

6. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to Event-Free Survival (EFS; Excluding SPNBC) Criteria
Description: Event-free survival (EFS) excluding second primary non-breast cancer (SPNBC) is defined as the time from enrollment to the first occurrence of one of the following events: breast cancer progression; breast cancer recurrence; or death from any cause. Ipsilateral or contralateral in situ disease and SPNBC (including in situ carcinomas and non-melanoma skin cancers) will not be counted as progressive disease or relapse.
Time Frame: At 1, 2, 3, and 4 years
Population: ITT Population. The number analyzed at each landmark timepoint represents the number of participants who were remaining at risk for an event.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Percentage of participants
  1 Year: number analyzed (Participants) | 237 | 235
  1 Year | 96.79 [94.60 to 98.98] | 97.95 [96.18 to 99.73]
  2 Years: number analyzed (Participants) | 224 | 218
  2 Years | 92.29 [88.96 to 95.62] | 91.67 [88.17 to 95.16]
  3 Years: number analyzed (Participants) | 212 | 209
  3 Years | 89.77 [85.96 to 93.57] | 88.29 [84.21 to 92.37]
  4 Years: number analyzed (Participants) | 191 | 198
  4 Years | 88.47 [84.44 to 92.49] | 86.57 [82.24 to 90.90]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only; p = 0.4844, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.72 to 1.98]

7. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to EFS (Including SPNBC) Criteria
Description: Event-free survival (EFS) including second primary non-breast cancer (SPNBC) is defined as the time from enrollment to the first occurrence of one of the following events: breast cancer progression; breast cancer recurrence; or death from any cause. It also includes SPNBC as an event (with the exception of non-melanoma skin cancers and in situ carcinoma of any site).
Time Frame: At 1, 2, 3, and 4 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Percentage of participants
  1 Year: number analyzed (Participants) | 236 | 234
  1 Year | 96.38 [94.06 to 98.70] | 97.54 [95.59 to 99.48]
  2 Years: number analyzed (Participants) | 222 | 215
  2 Years | 91.47 [87.98 to 94.96] | 90.41 [86.69 to 94.14]
  3 Years: number analyzed (Participants) | 209 | 206
  3 Years | 88.53 [84.52 to 92.53] | 87.04 [82.78 to 91.30]
  4 Years: number analyzed (Participants) | 188 | 196
  4 Years | 87.22 [83.02 to 91.43] | 85.75 [81.31 to 90.18]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only; p = 0.5474, Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.71 to 1.88]

8. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to Distant Recurrence-Free Interval (DRFI) Criteria
Description: The distant recurrence-free interval (DRFI) is defined as the time between randomization and the date of distant breast cancer recurrence.
Time Frame: At 1, 2, 3, and 4 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Percentage of participants
  1 Year: number analyzed (Participants) | 244 | 239
  1 Year | 99.59 [98.80 to 100.00] | 99.58 [98.77 to 100.00]
  2 Years: number analyzed (Participants) | 231 | 224
  2 Years | 95.88 [93.39 to 98.38] | 95.37 [92.70 to 98.04]
  3 Years: number analyzed (Participants) | 221 | 216
  3 Years | 93.77 [90.72 to 96.82] | 93.23 [90.02 to 96.43]
  4 Years: number analyzed (Participants) | 212 | 210
  4 Years | 92.49 [89.15 to 95.83] | 91.92 [88.44 to 95.41]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only; p = 0.6291, Log Rank; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.61 to 2.24]

9. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants in Overall Survival
Description: Overall survival is defined as the time from randomization to death from any cause.
Time Frame: At 1, 2, 3, and 4 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Percentage of participants
  1 Year: number analyzed (Participants) | 245 | 240
  1 Year | 99.60 [98.82 to 100.00] | 99.19 [98.06 to 100.00]
  2 Years: number analyzed (Participants) | 241 | 230
  2 Years | 98.38 [96.80 to 99.95] | 96.68 [94.42 to 98.94]
  3 Years: number analyzed (Participants) | 232 | 226
  3 Years | 96.73 [94.50 to 98.96] | 95.83 [93.30 to 98.36]
  4 Years: number analyzed (Participants) | 223 | 221
  4 Years | 95.47 [92.86 to 98.09] | 94.13 [91.14 to 97.11]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only; p = 0.5609, Log Rank; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.58 to 2.72]

10. Secondary Outcome: Summary of the Number of Participants With at Least One Adverse Event, Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0), Over the Course of the Entire Study
Description: The adverse event (AE) severity grading scale for the NCI CTCAE v4.0 was used for assessing AE severity. Any AEs that were not specifically listed in the NCI CTCAE, v4.0 were graded per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to AE. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: From first dose of study treatment until 28 days after last dose of study treatment (up to 1 year, 6 months)
Population: Safety Population: includes all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Participants
  Any Adverse Event (AE): Any Grade | 251 | 248
  AE with Fatal Outcome (Grade 5) | 2 | 2
  Any AE: Grades 3 to 5 | 149 | 132
  Serious AE | 52 | 49
  Related Serious AE | 29 | 29
  Anaphylaxis and Hypersensitivity AEs, Any Grade | 3 | 3
  Anaphylaxis and Hypersensitivity AEs, Grade ≥3 | 1 | 0
  Infusion/Admin.-Related Reactions Within 24 hrs, Any Grade | 39 | 54
  Infusion/Admin.-Related Reactions Within 24 hrs, Grade ≥3 | 3 | 0
  Serious Rash/Skin Reactions, Any Grade | 0 | 1
  Serious Rash/Skin Reactions, Grade ≥3 | 0 | 0
  Diarrhoea, Any Grade | 149 | 153
  Diarrhoea, Grade ≥3 | 13 | 16
  Cardiac Dysfunction, Any Grade | 65 | 52
  Cardiac Dysfunction, Grade ≥3 | 12 | 3
  Interstitial Lung Disease, Any Grade | 3 | 5
  Interstitial Lung Disease, Grade ≥3 | 0 | 0
  Neutropenia/Febrile Neutropenia, Any Grade | 142 | 123
  Neutropenia/Febrile Neutropenia, Grade ≥3 | 92 | 82
  Serious Mucositis, Any Grade | 3 | 3
  Serious Mucositis, Grade ≥3 | 3 | 2
  Pregnancy- and Neonatal-Related AEs, Any Grade | 0 | 0
  AE Leading to Study Drug Discontinuation | 32 | 22
  AE Leading to HER2-Targeted Therapy Discontinuation | 15 | 12
  AE Leading to Any Chemotherapy Drug Discontinuation | 23 | 14

11. Secondary Outcome: Number of Participants With a Primary Cardiac Event During the Neoadjuvant Phase
Description: A primary cardiac event is defined as the occurrence of either of the following events: - Incidence of a symptomatic ejection fraction decrease (heart failure) of New York Heart Association (NYHA) Class III or IV and a drop in left ventricular ejection fraction (LVEF) of at least 10-percentage points from baseline and to below 50%; or - Cardiac death, defined as: Definite cardiac death (due to heart failure, myocardial infarction, or documented primary arrhythmia); or, Probable cardiac death (sudden unexpected death within 24 hours of a definite or probable cardiac event [e.g., syncope, cardiac arrest, chest pain, infarction, arrhythmia] without documented etiology).
Time Frame: From first dose of study treatment until the completion of neoadjuvant therapy (24 weeks)
Population: Safety Population: includes all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Participants
  Any Primary Cardiac Event | 0 | 2
  Heart Failure and Significant LVEF Decline | 0 | 1
  Cardiac Death (Definite or Probable) | 0 | 1

12. Secondary Outcome: Number of Participants With a Secondary Cardiac Event During the Neoadjuvant Phase
Description: A secondary cardiac event is defined as asymptomatic or mildly symptomatic Left Ventricular Systolic Dysfunction (LVSD) of NYHA Class II, defined as a left ventricular ejection fraction (LVEF) decrease of at least 10-percentage points below the baseline measurement to an absolute LVEF value of <50% confirmed by a second assessment within approximately 3 weeks.
Time Frame: From first dose of study treatment until the completion of neoadjuvant therapy (24 weeks)
Population: Safety Population: includes all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Participants
  Any Secondary Cardiac Event | 4 | 1
  Identified by Initial LVEF Assessment | 4 | 1
  Confirmed by Second LVEF Assessment | 1 | 1

13. Secondary Outcome: Number of Participants With a Primary Cardiac Event During the Adjuvant Phase
Description: as for outcome 11
Time Frame: From surgery until 28 days after the last dose of adjuvant treatment (42 weeks)
Population: Safety Population: includes all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Participants
  Any Primary Cardiac Event | 1 | 2
  Heart Failure and Significant LVEF Decline | 1 | 2
  Cardiac Death (Definite or Probable) | 1 | 0

14. Secondary Outcome: Number of Participants With a Secondary Cardiac Event During the Adjuvant Phase
Description: as for outcome 12
Time Frame: From surgery until 28 days after the last dose of adjuvant treatment (42 weeks)
Population: Safety Population: includes all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Participants
  Any Secondary Cardiac Event | 15 | 8
  Identified by Initial LVEF Assessment | 15 | 8
  Confirmed by Second LVEF Assessment | 0 | 0

15. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities at the Highest NCI CTCAE v4 Grade Post-Baseline Over the Course of the Entire Study
Description: Clinical laboratory tests were performed at local laboratories; any abnormal values (High or Low) were based on local laboratory normal ranges. Laboratory abnormalities are presented by the highest (worst) severity grade (according to NCI-CTCAE v4.0) post-baseline. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a medical intervention or a change in concomitant therapy. For a participant with multiple post-baseline abnormalities, only the highest (worst) grade for a given laboratory test is reported. 'Any Grade' indicates the total number of participants with a post-baseline abnormality of any grade for the specified test.
Time Frame: From first dose of study treatment until 28 days after last dose of study treatment (up to 1 year, 6 months)
Population: Safety Population: includes all participants who received at least one dose of study medication. The number analyzed varies because it indicates all participants with a post-baseline laboratory value for a given test within the timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 252 | 248
Participants
  Albumin, Low - Any Grade: number analyzed (Participants) | 251 | 247
  Albumin, Low - Any Grade | 50 | 39
  Albumin, Low - Grade 1: number analyzed (Participants) | 251 | 247
  Albumin, Low - Grade 1 | 41 | 34
  Albumin, Low - Grade 2: number analyzed (Participants) | 251 | 247
  Albumin, Low - Grade 2 | 8 | 5
  Albumin, Low - Grade 3: number analyzed (Participants) | 251 | 247
  Albumin, Low - Grade 3 | 1 | 0
  Alkaline Phosphatase, High - Any Grade: number analyzed (Participants) | 234 | 225
  Alkaline Phosphatase, High - Any Grade | 80 | 71
  Alkaline Phosphatase, High - Grade 1: number analyzed (Participants) | 234 | 225
  Alkaline Phosphatase, High - Grade 1 | 78 | 70
  Alkaline Phosphatase, High - Grade 2: number analyzed (Participants) | 234 | 225
  Alkaline Phosphatase, High - Grade 2 | 2 | 1
  SGPT/ALT, High - Any Grade | 172 | 149
  SGPT/ALT, High - Grade 1 | 145 | 132
  SGPT/ALT, High - Grade 2 | 18 | 13
  SGPT/ALT, High - Grade 3 | 9 | 4
  SGOT/AST, High - Any Grade | 149 | 130
  SGOT/AST, High - Grade 1 | 137 | 125
  SGOT/AST, High - Grade 2 | 7 | 3
  SGOT/AST, High - Grade 3 | 5 | 2
  Creatinine, High - Any Grade | 225 | 217
  Creatinine, High - Grade 1 | 214 | 204
  Creatinine, High - Grade 2 | 9 | 13
  Creatinine, High - Grade 3 | 2 | 0
  Glucose, Low - Any Grade: number analyzed (Participants) | 251 | 247
  Glucose, Low - Any Grade | 23 | 22
  Glucose, Low - Grade 1: number analyzed (Participants) | 251 | 247
  Glucose, Low - Grade 1 | 20 | 22
  Glucose, Low - Grade 2: number analyzed (Participants) | 251 | 247
  Glucose, Low - Grade 2 | 3 | 0
  Glucose, High - Any Grade: number analyzed (Participants) | 251 | 247
  Glucose, High - Any Grade | 3 | 4
  Glucose, High - Grade 3: number analyzed (Participants) | 251 | 247
  Glucose, High - Grade 3 | 3 | 4
  Hemoglobin, Low - Any Grade | 233 | 223
  Hemoglobin, Low - Grade 1 | 129 | 139
  Hemoglobin, Low - Grade 2 | 93 | 77
  Hemoglobin, Low - Grade 3 | 11 | 7
  Hemoglobin, High - Any Grade | 12 | 6
  Hemoglobin, High - Grade 1 | 12 | 6
  Lymphocytes, Abs., Low - Any Grade: number analyzed (Participants) | 163 | 167
  Lymphocytes, Abs., Low - Any Grade | 144 | 150
  Lymphocytes, Abs., Low - Grade 1: number analyzed (Participants) | 163 | 167
  Lymphocytes, Abs., Low - Grade 1 | 23 | 22
  Lymphocytes, Abs., Low - Grade 2: number analyzed (Participants) | 163 | 167
  Lymphocytes, Abs., Low - Grade 2 | 59 | 68
  Lymphocytes, Abs., Low - Grade 3: number analyzed (Participants) | 163 | 167
  Lymphocytes, Abs., Low - Grade 3 | 55 | 56
  Lymphocytes, Abs., Low - Grade 4: number analyzed (Participants) | 163 | 167
  Lymphocytes, Abs., Low - Grade 4 | 7 | 4
  Lymphocytes, Abs., High - Any Grade: number analyzed (Participants) | 163 | 167
  Lymphocytes, Abs., High - Any Grade | 4 | 3
  Lymphocytes, Abs., High - Grade 2: number analyzed (Participants) | 163 | 167
  Lymphocytes, Abs., High - Grade 2 | 4 | 3
  Neutrophils, Total, Abs., Low - Any Grade: number analyzed (Participants) | 163 | 167
  Neutrophils, Total, Abs., Low - Any Grade | 110 | 114
  Neutrophils, Total, Abs., Low - Grade 1: number analyzed (Participants) | 163 | 167
  Neutrophils, Total, Abs., Low - Grade 1 | 27 | 42
  Neutrophils, Total, Abs., Low - Grade 2: number analyzed (Participants) | 163 | 167
  Neutrophils, Total, Abs., Low - Grade 2 | 30 | 23
  Neutrophils, Total, Abs., Low - Grade 3: number analyzed (Participants) | 163 | 167
  Neutrophils, Total, Abs., Low - Grade 3 | 17 | 24
  Neutrophils, Total, Abs., Low - Grade 4: number analyzed (Participants) | 163 | 167
  Neutrophils, Total, Abs., Low - Grade 4 | 36 | 25
  Platelets, Low - Any Grade | 72 | 67
  Platelets, Low - Grade 1 | 68 | 65
  Platelets, Low - Grade 2 | 3 | 2
  Platelets, Low - Grade 3 | 1 | 0
  Potassium, Low - Any Grade | 45 | 41
  Potassium, Low - Grade 2 | 38 | 28
  Potassium, Low - Grade 3 | 6 | 11
  Potassium, Low - Grade 4 | 1 | 2
  Potassium, High - Any Grade | 24 | 32
  Potassium, High - Grade 1 | 17 | 26
  Potassium, High - Grade 2 | 7 | 3
  Potassium, High - Grade 3 | 0 | 2
  Potassium, High - Grade 4 | 0 | 1
  Sodium, Low - Any Grade | 27 | 33
  Sodium, Low - Grade 1 | 22 | 32
  Sodium, Low - Grade 3 | 4 | 0
  Sodium, Low - Grade 4 | 1 | 1
  Sodium, High - Any Grade | 25 | 16
  Sodium, High - Grade 1 | 19 | 13
  Sodium, High - Grade 2 | 4 | 1
  Sodium, High - Grade 3 | 0 | 1
  Sodium, High - Grade 4 | 2 | 1
  Bilirubin, High - Any Grade | 24 | 22
  Bilirubin, High - Grade 1 | 16 | 17
  Bilirubin, High - Grade 2 | 7 | 5
  Bilirubin, High - Grade 3 | 1 | 0
  Total Leukocyte Count, Low - Any Grade | 199 | 203
  Total Leukocyte Count, Low - Grade 1 | 57 | 64
  Total Leukocyte Count, Low - Grade 2 | 81 | 78
  Total Leukocyte Count, Low - Grade 3 | 41 | 43
  Total Leukocyte Count, Low - Grade 4 | 20 | 18
  Total Leukocyte Count, High - Any Grade | 0 | 1
  Total Leukocyte Count, High - Grade 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs): From first dose of study treatment until 28 days after last dose of study treatment (up to 1 year, 6 months); All-cause mortality: From first dose of study treatment until end of follow-up (up to 4 years, 11 months)
Description: After initiation of study drug, all AEs were reported until 28 days after the last dose of study drug. After this period, only drug-related serious AEs, heart failure, pregnancies, and malignancies were reported.
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 12/252 | 14/248
Serious Adverse Events (participants affected / at risk) | 52/252 | 49/248
Other Adverse Events (participants affected / at risk) | 251/252 | 248/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy (N=252) | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy (N=248)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (11) | 9 (9)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 6 (6) | 4 (5)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Lithiasis (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 2 (2) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 3 (4)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flap necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy (N=252) | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy (N=248)
Anaemia (Blood and lymphatic system disorders) | 109 (148) | 90 (117)
Leukopenia (Blood and lymphatic system disorders) | 36 (58) | 25 (42)
Neutropenia (Blood and lymphatic system disorders) | 64 (119) | 58 (109)
Dry eye (Eye disorders) | 9 (11) | 14 (14)
Lacrimation increased (Eye disorders) | 14 (15) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 15 (17) | 22 (29)
Abdominal pain upper (Gastrointestinal disorders) | 21 (25) | 20 (31)
Constipation (Gastrointestinal disorders) | 54 (79) | 57 (75)
Diarrhoea (Gastrointestinal disorders) | 148 (309) | 152 (293)
Dyspepsia (Gastrointestinal disorders) | 31 (34) | 35 (42)
Gastritis (Gastrointestinal disorders) | 5 (6) | 13 (14)
Haemorrhoids (Gastrointestinal disorders) | 11 (11) | 22 (22)
Nausea (Gastrointestinal disorders) | 157 (327) | 151 (308)
Stomatitis (Gastrointestinal disorders) | 61 (90) | 63 (85)
Vomiting (Gastrointestinal disorders) | 50 (73) | 50 (71)
Asthenia (General disorders) | 84 (142) | 79 (160)
Fatigue (General disorders) | 62 (114) | 71 (113)
Influenza like illness (General disorders) | 11 (17) | 15 (21)
Injection site reaction (General disorders) | 2 (2) | 40 (174)
Malaise (General disorders) | 16 (20) | 14 (20)
Mucosal inflammation (General disorders) | 49 (66) | 39 (53)
Oedema (General disorders) | 13 (13) | 6 (6)
Oedema peripheral (General disorders) | 26 (28) | 23 (25)
Pyrexia (General disorders) | 41 (56) | 32 (41)
Cystitis (Infections and infestations) | 13 (14) | 8 (8)
Nasopharyngitis (Infections and infestations) | 36 (39) | 33 (40)
Paronychia (Infections and infestations) | 12 (14) | 20 (21)
Rhinitis (Infections and infestations) | 13 (17) | 14 (15)
Upper respiratory tract infection (Infections and infestations) | 24 (37) | 34 (43)
Urinary tract infection (Infections and infestations) | 16 (20) | 18 (22)
Infusion related reaction (Injury, poisoning and procedural complications) | 36 (53) | 9 (9)
Procedural pain (Injury, poisoning and procedural complications) | 25 (26) | 29 (31)
Radiation skin injury (Injury, poisoning and procedural complications) | 54 (55) | 50 (51)
Alanine aminotransferase increased (Investigations) | 50 (61) | 39 (50)
Aspartate aminotransferase increased (Investigations) | 40 (54) | 29 (37)
Ejection fraction decreased (Investigations) | 24 (28) | 16 (17)
Neutrophil count decreased (Investigations) | 54 (141) | 40 (97)
Weight decreased (Investigations) | 15 (16) | 26 (27)
White blood cell count decreased (Investigations) | 35 (108) | 19 (58)
Decreased appetite (Metabolism and nutrition disorders) | 51 (70) | 43 (50)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (24) | 16 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 (106) | 71 (91)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (20) | 25 (32)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (19) | 20 (24)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 (20) | 21 (23)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (18) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 52 (63) | 67 (80)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (30) | 22 (26)
Dizziness (Nervous system disorders) | 32 (39) | 34 (39)
Dysgeusia (Nervous system disorders) | 35 (45) | 43 (53)
Headache (Nervous system disorders) | 68 (84) | 45 (72)
Neuropathy peripheral (Nervous system disorders) | 40 (53) | 33 (38)
Paraesthesia (Nervous system disorders) | 23 (26) | 25 (30)
Peripheral sensory neuropathy (Nervous system disorders) | 40 (44) | 42 (45)
Anxiety (Psychiatric disorders) | 8 (8) | 15 (17)
Insomnia (Psychiatric disorders) | 35 (45) | 44 (50)
Breast pain (Reproductive system and breast disorders) | 13 (13) | 15 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (43) | 41 (44)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 29 (32)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 37 (43) | 31 (36)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (21) | 15 (16)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 17 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 184 (188) | 196 (196)
Dermatitis (Skin and subcutaneous tissue disorders) | 14 (14) | 19 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 34 (39) | 38 (43)
Erythema (Skin and subcutaneous tissue disorders) | 14 (14) | 22 (26)
Nail discolouration (Skin and subcutaneous tissue disorders) | 17 (17) | 23 (23)
Nail disorder (Skin and subcutaneous tissue disorders) | 17 (17) | 16 (18)
Onycholysis (Skin and subcutaneous tissue disorders) | 13 (13) | 11 (11)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 (13) | 17 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (29) | 29 (35)
Rash (Skin and subcutaneous tissue disorders) | 56 (75) | 46 (56)
Hot flush (Vascular disorders) | 39 (44) | 41 (44)
Hypertension (Vascular disorders) | 16 (19) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03493854/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT03493854/SAP_001.pdf